CLINICAL TRIAL: NCT01876849
Title: An Open-Label Study Examining the Long-Term Safety of Exenatide Given Twice Daily to Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H8O-MC-GWAN
Record Dates: First submitted 2009-07-14; First posted 2013-06-13 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide; Byetta; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group A (Experimental): Exenatide injection 5mcg or 10 mcg, twice daily
  Interventions: Drug: exenatide

INTERVENTIONS:
Drug: exenatide — subcutaneous injection, 5mcg or 10 mcg, twice daily
  Other Names: Byetta

SUMMARY:
The aim of this study is to assess the long-term safety of exenatide in patients with type 2 diabetes who were treated with exenatide in Study H8O-MC-GWAA (6-month study) or Study H8O-MC-GWAD (12-month study). Study H8O-MC-GWAN serves as an open-ended extension to Studies H8O-MC-GWAA and H8O-MC-GWAD.

ELIGIBILITY:
Inclusion Criteria:

* Patients received exenatide therapy in Study H8O-MC-GWAA or Study H8O-MC-GWAD and completed the respective study.

Exclusion Criteria:

* Patients were excluded or discontinued early from Study H8O-MC-GWAA or Study H8O-MC-GWAD.
* Patients have received treatment within the last 30 days with a drug, not including exenatide, that has not received regulatory approval for any indication at the time of study entry.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2003-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Long-term safety of twice-daily exenatide treatment, as defined by the occurrence of adverse events. | 128 weeks (average treatment period)
  Visits for this study occur at 6-mo (±2 wk) intervals until exenatide is approved for marketing.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, MD, Study Director — Eli Lilly and Company
Locations (1):
- Research Site, Renton, Washington, United States